CLINICAL TRIAL: NCT01461720
Title: An Open Lable, Phase II Exploratory Study Assessing the Efficacy of Intravenous Autologous Mesenchymal Stem Cells in Patients With Middle Cerebral Artery Infarct
Brief Title: Intravenous Autologous Mesenchymal Stem Cells Transplantation to Treat Middle Cerebral Artery Infarct
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Cytopeutics Sdn. Bhd. (Industry)
Responsible Party: Principal Investigator, Dr Norlinah Mohamed Ibrahim, Consultant Neurologist, National University of Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF-115-2011
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Middle Cerebral Artery Infarction
Keywords: Bone marrow; Autologous; Mesenchymal stem cells; Unilateral middle cerebral artery infarct
MeSH Terms: conditions — Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard medical care (Other): This is the control arm, which is given the best evidence-based standard treatment for the management of acute stroke
  Interventions: Other: Standard medical care
- BM-MSCs (Experimental): Autologous bone marrow-derived mesenchymal stem cells(BM-MSCs)
  Interventions: Other: Standard medical care; Biological: Autologous bone marrow-derived mesenchymal stem cells

INTERVENTIONS:
Other: Standard medical care — Standard medical care includes treatment to prevent recurrence, optimal control of risk factors and post stroke follow-up rehabilitative treatment.
Biological: Autologous bone marrow-derived mesenchymal stem cells — Single intravenous infusion of autologous bone marrow-derived mesenchymal stem cells concurrently with standard medical care.
  Arms: BM-MSCs

SUMMARY:
This study aims to determine the efficacy of intravenous transplantation of autologous bone marrow-derived mesenchymal stem cells in patients with acute middle cerebral artery infarct.

ELIGIBILITY:
Inclusion Criteria:

* Experiences stroke onset within 2 weeks to 2 months
* NIHSS score of >10-35
* Never received or failed thrombolysis
* Evidence of unilateral middle cerebral artery infarct on brain MRI

Exclusion Criteria:

* Medically unfit (eg. those are unstable haemodynamically despite treatment, with worsening conscious level and with other serious medical co-morbidity)
* Evidence of any tumor or other space-occupying lesion on brain MRI
* Evidence of hemorrhagic stroke on brain CT or MRI
* Experiences transient ischemic attack or lacunar infarct
* Has any acute or chronic infections such as Hepatitis B, Hepatitis C and HIV
* Is diagnosed with concurrent malignancy or primary hematological disorders
* Renal impairment indicated with serum creatinine greater than 200 umol/l or creatinine clearance less than 30 ml/min
* Liver impairment indicated with serum aspartate transaminase and serum alanine transaminase greater than 4 times upper limit of the normal range
* Any contraindication to stem cell transplantation or bone marrow biopsy
* Any co-morbidity which will compromise the ability to obtain adequate stem cells (eg. chronic debilitating diseases, frail patients and patients with known osteoporosis)
* Any contraindication to brain MRI (eg. metal implants, pacemaker, joint implants and ocular implants)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in NIH Stroke Scale | 1 year
Change in Barthel Index | 1 year
Change in modified Rankin Scale | 1 year
Change in size of infarct based on brain MRI stroke sequences | 1 year

SECONDARY OUTCOMES:
Change in Stroke Specific Quality of Life Scale | 1 year
Change in Stroke Impact Scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Norlinah Mohamed Ibrahim, MD, Principal Investigator — UKM Medical Centre
Locations (1):
- UKM Medical Centre, Kuala Lumpur, Malaysia